CLINICAL TRIAL: NCT06646341
Title: EMVI as a Determinant of Metastasis in Colorectal Cancer
Acronym: EVIDENCE
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: DOCUMAS: 22HH7583
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Colo-rectal Cancer
Keywords: Extramural Venous Invasion; Extranodal Tumour Deposits; Imaging and Pathology Biomarkers; Pelvic Recurrence; Colorectal Cancer; Local Advanced Rectal Cancer; Metastatic Spread; MRI staging; Phylogenesis; Rectal Cancer Recurrence; Sigmoid Cancer; Surgery for Pelvic Recurrence
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms; Sigmoid Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Biopsy and resection specimens: Formalin-Fixed Paraffin-Embedded (FFPE) tissue blocks, (Hematoxylin and Eosin) H&E slides, High resolution digital slides
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Bowel cancer is the fourth most commonly occurring cancer and the second highest cause of cancer deaths in the UK. Despite advances in treatment, over 40% of patients will die within 5 years. This is normally due to spread of the cancer to other organs (called metastases). Much of the current research focuses on use of additional treatments such as radiotherapy and chemotherapy before or after surgery (adjuvant treatment). It is of vital importance that patients who would benefit from adjuvant treatment can be accurately identified. At the moment, the system used locally to do this places emphasis on the presence of affected lymph nodes (glands). This is because doctors believe that cancer spreads to other organs through the lymphatic system. However, recent studies have suggested that this is not the case.

It is believed that cancer spreads to other organs through the blood stream rather than the lymph node system. This research will look at the genetic material in tumours and metastases as well as in areas of blood vessel invasion and lymph nodes. The analysis will allow us to build a 'family tree' of the tumour and allow us to map the pathway by which the tumour spreads. Tissue samples already collected through a patient's routine care will be used for this study. If the spread through the blood vessels is proven, this would change the way in which patients are selected for treatment and allow development of new treatments to target these pathways.

DETAILED DESCRIPTION:
A retrospective ,non-interventional tissue study using archival materials collected through a patient's routine care, EVIDENCE aims to demonstrate that distant metastases in colorectal cancer are related to Extramural Venous Invasion (EMVI) and tumour deposits, not lymph nodes. As EVIDENCE is a retrospective study, there are no time dependent schedules for Case Report Form (CRF) completion or tissue submission.

It will be tested whether the vascular route of spread (as evidenced through EMVI and tumour deposits) is more important than lymph nodes in the development of metastatic disease. The sub-clonal origins of primary colorectal cancers, EMVI, tumour deposits, lymph nodes and distant metastases by reconstructing phylogenetic trees will be compared. A proof for a vascular route of spread rather than lymph nodes would lead to a paradigm shift in future decision making at national and international level.

ELIGIBILITY:
Inclusion Criteria:

1. Are aged 16 years or over with colorectal cancer
2. Colon / rectum has been surgically removed
3. Distant metastases has been surgically removed
4. Pre operative staging in the form of CT/MRI has been undertaken and images available for review

Exclusion Criteria:

1. Pathological complete response in the primary tumour
2. Local resection of the primary tumour
3. Inadequate quantity of tissue sample to perform analyses

Ages: 16 Years to 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have undergone a primary resection of their colon or rectum as well as a resection of a distant metastases
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of proportion of subjects where Extramural Venous Invasion (EMVI) and tumour deposits vs lymph nodes are associated with distant metastases | 1 year from last registered patient
  Proportion of subjects where EMVI and tumour deposits rather than lymph nodes are associated with distant metastases. This is to determine the route of spread of distant metastases.

SECONDARY OUTCOMES:
Comparison of tumour phylogenetic profile between primary tumour, EMVI, tumour deposits, metastases | 1 year from last registered patient
  Comparison of tumour phylogenetic profile between primary tumour, EMVI, tumour deposits, metastases. This is to investigate the clonal origins of metastases in relation to the primary tumour deposits, EMVI and lymph nodes
Comparison of tumour phylogenes between different metastatic sites and primary tumour | 1 year from last registered patient
  Comparison of tumour phylogenes between different metastatic sites and primary tumour. This is to determine if there are different routes of spread to different organs (i.e. lung, liver, brain, peritoneal)
Comparison of immunohistochemistry staining profile between primary tumour, EMVI, tumour deposits, metastases | 1 year from last registered patient
  Comparison of immunohistochemistry staining profile between primary tumour, EMVI, tumour deposits, metastases. This is to evaluate the similarities in the immunohistochemistry profile of metastases compared with primary tumour deposits, EMVI and lymph nodes
Comparison of overall survival based on clonal origins of metastases | 1 year from last registered patient
  Comparison of overall survival based on clonal origins of metastases. This is to investigate the relationship between the clonal origins of metastases and outcomes according to primary tumour deposits, EMVI and lymph nodes

CONTACTS AND LOCATIONS:
Overall Officials: Gina Brown, MD, Principal Investigator — Imperial College London
Locations (1):
- Hampshire Hospitals Nhs Foundation Trust, Basingstoke, Hampshire, United Kingdom